CLINICAL TRIAL: NCT01789411
Title: The European Collaborative Project on Inflammation and Vascular Wall Remodeling in Atherosclerosis - Intravascular Ultrasound Study
Acronym: AtheroRemoIVUS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Patrick W. Serruys, MD, PhD, Erasmus Medical Center
Other Study IDs: EMC MEC 2008-210
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ATHEROREMO-IVUS cohort: Drawing blood samples. Coronary intravascular ultrasound imaging. Coronary near-infrared spectroscopy.
  Interventions: Other: Drawing blood samples; Device: Coronary intravascular ultrasound imaging; Device: Coronary near-infrared spectroscopy

INTERVENTIONS:
Other: Drawing blood samples — Drawing blood samples from the arterial sheath prior to the standard coronary angiography procedure
Device: Coronary intravascular ultrasound imaging — Coronary intravascular ultrasound imaging of a non-culprit coronary artery.
Device: Coronary near-infrared spectroscopy — Near-infrared spectroscopy imaging of a non-culprit coronary artery (in patient who are included in the AtheroRemo-NIRS substudy).

SUMMARY:
The AtheroRemo-IVUS study aims to investigate the relation of coronary plaque phenotype and vulnerability as determined by intravascular ultrasound and near infrared spectroscopy with genetic profile and novel circulating biomarkers. AtheroRemo-IVUS is a prospective, observational, cohort study of patients who underwent coronary catheterization for acute coronary syndrome or stable angina pectoris. Prior to the catheterization procedure, blood samples were drawn for biomarker measurements and genetic analyses. Subsequent to the catheterization procedure, intravascular ultrasound is performed in a non-culprit coronary artery. In patients who are also participating in the AtheroRemo-NIRS substudy, near-infrared spectroscopy is additionally performed in the same non-culprit vessel. Primary endpoint is the presence of vulnerable plaque as determined by intravascular ultrasound. Secondary endpoint is long-term incidence of major adverse cardiac events. Results from AtheroRemo-IVUS are expected to improve our knowledge on the role of genetic profile and inflammation in the development of atherosclerosis and vulnerable plaques. Furthermore, novel biomarkers and intracoronary imaging techniques will be validated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, more than 21 years old.
2. Patients with stable angina pectoris (CCS Class 1, 2, 3 or 4) or unstable angina pectoris (Braunwald Class 1-3, B-C) or patients with documented silent ischemia or patients with an acute myocardial infarction (STEMI and NSTEMI).
3. Patients eligible for coronary revascularization in the native coronary artery/arteries.
4. Willing and able to comply with the specified follow-up evaluation.
5. Written informed consent obtained.
6. Flow-limiting stenosis (diameter stenosis ≥50% by QCA or visual estimate) that is held responsible for angina pectoris or acute coronary syndrome
7. The study vessel has not undergone percutaneous coronary intervention in the last 8 months.

Exclusion Criteria:

1. Braunwald class IA, IIA, IIIA (angina caused by non-cardiac illness).
2. Women who are pregnant or women of childbearing potential who do not use adequate contraception.
3. Known allergies to aspirin, clopidogrel bisulfate (Plavix ®), Ticlopdine (Ticlid ®) heparin, stainless steel, copper or a sensitivity to contrast media which cannot be adequately pre-medicated.
4. Previous participation in this study or participation in another study with any investigational drug or device within the past 30 days (study participation ends after completion of the final follow-up.)
5. Life expectancy of less than one year or factors making clinical and/or angiographic follow-up difficult.
6. Planned or being status post coronary bypass surgery.
7. Planned major non-cardiac surgery.
8. Impaired renal function (creatinine >2 mg/dl or >150 umol/L).
9. The subject has a history of bleeding diathesis or coagulopathy.
10. The subject suffered disabling stroke within the past year.
11. 3-vessel coronary artery and/or Left main disease with > 50% stenosis.
12. Minimal lumen diameter <2mm in the segments to be analyzed within the study vessel.
13. Diameter Stenosis >70% or total occlusion of the study vessel.
14. In case the study-vessel has been stented previously (>8 months ago), more than 1/3 proximal of the study vessel (at least 40mm in length) should be available for examination (i.e., outside the length of the stent plus 5mm proximal to the stent).
15. Poor LV function as assessed by Echo or by Angiography.
16. The proximal vessel is moderately to severely tortuous (moderate: 2 bends >75 degrees or one bend >90 degrees) in the segment(s) to be analyzed.
17. Known tendency to coronary vasospasm.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome or stable angina pectoris, referred for percutaneous coronary intervention or coronary angiography
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Vulnerable plaque as determined by intravascular ultrasound | cross-sectional (time of baseline coronary angiography, no follow-up)
  The primary objective is to correlate coronary plaque phenotype as determined by intravascular ultrasound with genetic profile and circulating biomarkers. Primary endpoint is the presence of vulnerable plaque as determined by intravascular ultrasound.

SECONDARY OUTCOMES:
Major adverse cardiac events | 1-year follow-up
  The secondary objective is to assess the prognostic value of novel biomarkers and plaque phenotypes as determined by intravascular ultrasound and near-infrared spectroscopy. Secondary endpoint is 1-year incidence of major adverse cardiac events.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Derived] Schuurman AS, Vroegindewey MM, Kardys I, Oemrawsingh RM, Garcia-Garcia HM, van Geuns RJ, Regar E, Van Mieghem NM, Ligthart J, Serruys PW, Boersma E, Akkerhuis KM. Prognostic Value of Intravascular Ultrasound in Patients With Coronary Artery Disease. J Am Coll Cardiol. 2018 Oct 23;72(17):2003-2011. doi: 10.1016/j.jacc.2018.08.2140. PMID 30336823
- [Derived] de Boer S, Baran Y, Garcia-Garcia HM, Eskin I, Lenzen MJ, Kleber ME, Regar E, de Jaegere PJ, Ligthart JM, van Geuns RJ, Lehtimaki T, Laaksonen R, Boersma E, Marz W, Halperin E, Serruys PW, Koenig W. The European Collaborative Project on Inflammation and Vascular Wall Remodeling in Atherosclerosis - Intravascular Ultrasound (ATHEROREMO-IVUS) study. EuroIntervention. 2018 Jun 20;14(2):194-203. doi: 10.4244/EIJ-D-17-00180. PMID 28943493
- [Derived] Oemrawsingh RM, Cheng JM, Garcia-Garcia HM, van Geuns RJ, de Boer SP, Simsek C, Kardys I, Lenzen MJ, van Domburg RT, Regar E, Serruys PW, Akkerhuis KM, Boersma E; ATHEROREMO-NIRS Investigators. Near-infrared spectroscopy predicts cardiovascular outcome in patients with coronary artery disease. J Am Coll Cardiol. 2014 Dec 16;64(23):2510-8. doi: 10.1016/j.jacc.2014.07.998. PMID 25500237
- [Derived] Sonneveld MA, Cheng JM, Oemrawsingh RM, de Maat MP, Kardys I, Garcia-Garcia HM, van Geuns RJ, Regar E, Serruys PW, Boersma E, Akkerhuis KM, Leebeek FW. Von Willebrand factor in relation to coronary plaque characteristics and cardiovascular outcome. Results of the ATHEROREMO-IVUS study. Thromb Haemost. 2015 Mar;113(3):577-84. doi: 10.1160/TH14-07-0589. Epub 2014 Dec 4. PMID 25472874
- [Derived] Cheng JM, Oemrawsingh RM, Akkerhuis KM, Garcia-Garcia HM, de Boer SP, Battes LC, Buljubasic N, Lenzen MJ, de Jaegere PP, van Geuns RJ, Serruys PW, Kardys I, Boersma E. Circulating chemokines in relation to coronary plaque characteristics on radiofrequency intravascular ultrasound and cardiovascular outcome. Biomarkers. 2014 Nov;19(7):611-9. doi: 10.3109/1354750X.2014.957725. Epub 2014 Sep 8. PMID 25196123
- [Derived] de Boer SP, Cheng JM, Garcia-Garcia HM, Oemrawsingh RM, van Geuns RJ, Regar E, Zijlstra F, Laaksonen R, Halperin E, Kleber ME, Koenig W, Boersma E, Serruys PW. Relation of genetic profile and novel circulating biomarkers with coronary plaque phenotype as determined by intravascular ultrasound: rationale and design of the ATHEROREMO-IVUS study. EuroIntervention. 2014 Dec;10(8):953-60. doi: 10.4244/EIJY13M08_01. PMID 24063848